CLINICAL TRIAL: NCT06384495
Title: How Does Cerebellar tDCS Alter Intracortical Inhibition Over Time?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. The duration of research tasks exceeded the expected timeframe for uncompensated participants
  2. The tDCS system was discontinued and therefore no longer serviced by the manufacturer.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00021475
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real anodal tDCS group (REAL-A) (Experimental): Participants randomized to REAL-A
  Interventions: Procedure: REAL-A
- Real cathodal tDCS group (REAL-C) (Experimental): Participants randomized to REAL-C
  Interventions: Procedure: REAL-C
- Sham group (SHAM) (Sham Comparator): Participants randomized to SHAM group
  Interventions: Procedure: SHAM

INTERVENTIONS:
Procedure: REAL-A — one session of 2mA for 20 minutes to the right ventro-lateral cerebellum
  Arms: Real anodal tDCS group (REAL-A)
Procedure: REAL-C — one session of 2mA for 20 minutes to the right ventro-lateral cerebellum
  Arms: Real cathodal tDCS group (REAL-C)
Procedure: SHAM — one session of sham tDCS for 20 minutes to the right ventro-lateral cerebellum.
  Arms: Sham group (SHAM)

SUMMARY:
Combining cortical tDCS with behavioral interventions has been shown to have beneficial outcomes in individuals post-stroke. However, cerebellar tDCS is a fairly new approach for individuals with unilateral cortical stroke and there has not been reports of duration of effect of tDCS applied to the cerebellum in this population.

Information gained from this study will serve to fill knowledge gaps on the duration of effect of cerebellar tDCS and the effects of polarity.

The purpose of this study is to determine the duration of effect of ventro-lateral cerebellar transcranial direct current stimulation (tDCS) in healthy adults through cortical excitability (CE), cognitive, language and motor assessment measures. Primary aim: Compare baseline CE from left motor cortex of first dorsal interosseous (FDI) and orbicularis oris (OO) areas to CE post cerebellar tDCS at 15 minutes, 45 minutes and 75 minutes. Single-pulse and paired-pulse transcranial magnetic stimulation (TMS) will be used to measure and compare stimulus response curve (S/R curve), cortical silent period (CSP) and short-interval intracortical inhibition (SICI) in the hand area and facial area of the left primary motor cortex at each time point.

Secondary aim: Compare baseline performance on cognition, motor learning and language tasks to performance at 15, 45 and 75 minutes after receiving tDCS. Digit Symbol Substitution Test (DSST), Serial Reaction Time Test (SRTT) and Lexical Decision tasks will be presented via a computer interface.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must be over the age of 18 years of age
* must be fluent in English
* have adequate vision to see a computer screen from 12-18 inches, fine motor skills to press a key on a computer keyboard and hearing to hear directions and questions provided by the researcher
* Individuals must also be able to read words and phrases

Exclusion Criteria:

* Pregnancy
* history of seizures
* neurologic injury including concussion/head injury or stroke or other neurologic conditions
* History of documented learning disabilities and/or ADHD
* Metal implants in the body (excluding dental fillings), psoriasis or eczema affecting the scalp.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
stimulus/response curve (S/R Curve) | baseline, 15,45 and 75 minutes post-tDCS
  change of motor evoked potential (MEP) as reflected in EMG from 1) hand (FDI muscle) and 2) mouth (orbicularis oris muscle).following single pulse transcranial magnetic stimulation (TMS) to the primary motor cortex of varying intensities.
Cortical Silent Period (CSP) | baseline, 15,45 and 75 minutes post-tDCS
  Change in silent period of a contracted muscle shown through EMG from 1) hand (FDI muscle) and 2) mouth (orbicularis oris muscle). following a single supra-threshold stimulus pulse to the primary motor cortex using TMS.
Short-interval Intracortical Inhibition (SICI). | baseline, 15,45 and 75 minutes post-tDCS
  Change in MEP as reflected in EMG from 1) hand (FDI muscle) and 2) mouth (orbicularis oris muscle). following a subthreshold conditioning pulse followed by a suprathreshold test pulse

SECONDARY OUTCOMES:
Digit Symbol Substitution Test (DSST) | baseline, 15, 45 and 75 minutes post stimulation
  The DSST is a 90-second timed test that evaluates processing speed, working memory, visuospatial processing, and attention. The test involves a subject replacing given numerals (1-9) with the corresponding unique, simple to draw, symbols provided in the key. The subject is instructed to write as many substitutions as possible within the allotted time. The score is determined by counting the correct number of substitutions. No penalty is applied for incorrect answers. The test permits freedom to achieve the task which allows for creativity and refinement to improve one's score. This test was originally a subsection of the Wechsler Adult Intelligence Test (WAIS), used to measure one's intelligence quotient (IQ)
Serial Reaction Time Test (SRTT) | baseline, 15, 45 and 75 minutes post stimulation
  The SRTT is a four-choice reaction time task that measures motor learning. In this task, a visual cue can appear at any one of four positions arranged horizontally on a computer screen. Each screen position, designated 1-4, corresponds to a button on a response pad. When a cue appears, at the start of each trial, a participant selects the appropriate response button. The visual cues play out a repeating sequence of positions (for example, 2-3-1-4-3-2-4-1-3-4-2-1). Sequential trials are followed by random trials
Lexical Decision Task | baseline, 15, 45 and 75 minutes post stimulation
  The lexical decision task requires the participant to make a decision whether a target letter string is a word or, with equal probability, a pronounceable non-word. The target string is preceded by a prime word that is either associated with the target word or, with equal probability, not associated

CONTACTS AND LOCATIONS:
Overall Officials: Sharyl Samargia-Grivette, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States